CLINICAL TRIAL: NCT05887856
Title: Reduction of Pre-operative Anxiety Using a Specially Designed Educational Program for Breast Cancer Patients Undergoing Surgery: a Randomized Controlled Trial
Acronym: PAUSDE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Awais Kanwal, Dr. Muhammad Awais Kanwal, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-22-40
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Patient Satisfaction; Preoperative Anxiety; Anxiety
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pre-operative randomization after enrollment will be carried out and patients will be allocated either to the "intervention group" or to the "non-intervention group "by 'computerized block randomization'. Research Randomizer software, a free to use software will be used for this. Patients will be randomized either into the intervention group or into non-intervention group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: It would be a "single blinded study" the assessor will be blinded to the type of group to which patient belongs.
  Blinding will be ensured by sharing the data only with relevant study team members, The assessor will read out instruction before beginning of the interview requesting the enrolled patients not to mention the tools used for pre-operative education and to answer only the questions being asked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Volunteers in the Intervention group will receive specially designed educational program which will be aimed at reduction of pre-operative anxiety in breast cancer patients undergoing surgery as a part of their treatment.
  Interventions: Other: comprehensive educational program for reduction of Pre-Operative Anxiety
- Non-Intervention Group (No Intervention): Non-Intervention group will get the usual standard information as per existing protocols which includes
  1. Explanation of surgical procedure by primary team.
  2. Information about anesthesia on pre-operative anesthesia assessment.
  3. Phone call from Primary team explaining surgery details one day prior to surgery in case of day case surgery.
  4. Information about surgery on admission from floor resident in case of Pre-Op Admission.
  Afore mentioned practices are standard at SKMCH and RC and will remain same for both intervention and non-intervention group.

INTERVENTIONS:
Other: comprehensive educational program for reduction of Pre-Operative Anxiety — BSEP 1 makes use of modern media and aims to educate patients and their carers through educational videos comprising of various aspect of surgical treatment.
  1. Introduction to surgery by consultant surgeon, Patient to receive video of their own surgeon.
  2. Introduction to Anesthesia.
  3. What are different type of breast surgeries in cancer patients (General Video)
  4. Specific video pertaining to the type of surgery patient is undergoing (Mastectomy, Breast Conserving Surgery, Breast Re Construction surgery)
  5. Explanation of Methicillin-resistant Staphylococcus aureus Decolonization protocol
  6. What to expect on Surgery Day
  7. Virtual tour of Holding bay and Operation Room
  8. Post-Operative care including wound care, drain management and common post-operative complications.
  Other Names: Breast Surgery Education Package 1 (BSEP 1)
  Arms: Intervention Group

SUMMARY:
This study aims to find out that if a specially designed educational program can help in reduction of pre-operative anxiety in breast cancer patients undergoing surgery as a part of their treatment.

DETAILED DESCRIPTION:
Anxiety can be defined as an unpleasant subjective experience associated with the perception of real threat; therefore, it is a common symptom in connection with cancer. Breast Cancer patients undergo surgery at some stage of their treatment, Surgery details can be overwhelming and might lead to low retention of information and greater levels of anxiety which is the most prevalent psychological symptoms perceived by cancer patients.

Studies have shown women with a diagnosis of cancer correlate with higher levels of preoperative anxiety. Increased anxiety elicits physiologic stress responses that may impede healing and alter responses to postoperative pain.It can also lead to delayed recovery, prolonged hospital stay and increased need of postoperative pain medications.

Pre-Operative Anxiety may also cause delayed recovery from Anesthesia and can also compromise the effectiveness of anesthesia .Furthermore, it can lead to other post-operative complications such as nausea, vomiting, and delayed wound healing. Various Pharmacological and non-pharmacological methods have been used for reduction of pre-operative anxiety and one such non-pharmacological method is educating the patients about the experience of surgery pre-operatively which we aim to study in our population.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years of age.
2. Known cases of Breast Cancer.
3. Undergoing Breast Surgery as a part of treatment.
4. Availability of Personal smart phone at home.
5. Written informed Consent given for participation in trial.
6. Females.

Exclusion Criteria:

1. Less than 18 years or more than 70 years of age.
2. Stage IV patients undergoing palliative breast surgery.
3. Patient having chronic pain.
4. Un-availability of smart phone.
5. Patients with known psychiatric/depression disorders.
6. Previous history of another treated carcinoma.
7. Patients with re-current breast carcinoma.
8. Male Patients are excluded from study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Patient Pre-Operative Anxiety | 6 months
  This will be measured by using The Perioperative Anxiety Scale-7 (PAS-7), PAS 7 is a validated tool which includes seven items. This tool was developed by Zhang, C., Liu, X., Hu, T. et al. at Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, China.
  Permissions were obtained and granted for use of PAS 7 in this project and its translation into Urdu. The process of translation involved forward translation by two independent translators, formation of a reconciled version by third translator, Back translation, independent review and finalization.

SECONDARY OUTCOMES:
Patient Satisfaction. | 6 Months
  This will be measured using Patient satisfaction questionnaire Short Form (PSQ-18). The short-form instrument, the PSQ-18, contains 18 items comprising of General satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, accessibility and convenience. PSQ-18 is a free to use validated tool developed by RAND Corporation. The translation of the tool is allowed by the RAND Corporation with precise instructions regarding the translation process. These instructions were followed while translating the tool. The process of translation involved forward translation by two independent translators, formation of a reconciled version by third translator, Back translation, independent review and finalization.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Barka Sajjad, M.B.B.S, FCPS, MRCS, Principal Investigator — Shaukat Khanum memorial cancer hospital and research centre lahore
Locations (1):
- Shaukat Khanum memorial cancer hospital and research centre, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No